CLINICAL TRIAL: NCT01407653
Title: Evaluation of the Analgesic Effect of a Prototype Device of Virtual Reality in a Population of Patients With Chronic Low Back Pain. A Randomized Controlled Trial Using a Modified ZELEN Method
Brief Title: Analgesic Effect of a Prototype Device of Virtual Reality in a Population of Patients With Chronic Low Back Pain
Acronym: REVLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: NEUROVIRTUAL (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P100302
Record Dates: First submitted 2011-05-30; First posted 2011-08-02 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; virtual reality
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- virtual reality (Experimental)
  Interventions: Procedure: Virtual reality
- usual care (Other)
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Virtual reality — 3 sessions of immersion in a virtual reality 3D environment of 17 minutes per week for 4 consecutive weeks
  Arms: virtual reality
Procedure: Usual care — Classical care
  Arms: usual care

SUMMARY:
Chronic low back pain and sciatica in adults represent a major medical and economic problem. During the chronic back pain (persisting continuously over 3 months), therapeutic responses to conventional pharmacologic type are often ineffective and the impact of pain is often heavy in terms of disability, social and professional avulsion and loss of quality of life. This failure has led in recent years to propose innovative strategies such as application of relaxation therapy techniques. An example is a virtual reality which is a technology to immerse someone in a 3D virtual environment. Our hypothesis is that the hypnotic suggestion combined with virtual reality can be effective on chronic pain. The main purpose is to measure the impact on the intensity of pain at 4 months after using of a new method for virtual environment, mimicking the colors from low to high frequencies (World Patent Filed, WO2007/057601) in patients with chronic disabling low back pain and sciatica resistant to therapeutic drugs.

DETAILED DESCRIPTION:
Secondary objectives:

* Quantifying the effects in terms of disability associated with chronic pain
* Quantifying the effects on the cognitive (affect, anxiety, depression).
* Study the correlation between pain and oxidative stress.

Methods :a controlled, randomized single-center prospective trial, according to a ZELEN modified scheme

Intervention treatment : Pain treatment by a process of Virtual Reality 3D. The intervention protocol consists of 3 sessions of immersion in a 3D environment of 17 minutes per week for 4 consecutive weeks.

Conducting the study: an inclusion visit, then the intervention protocol for patients in the arm "Virtual Reality" during 4 weeks, and then a monthly follow-up visit for 4 months.

V0 - Inclusion Visit

* Physical examination
* Verification of eligibility
* Proposal of the trial cohort and collection of the informed consent, signed
* Inclusion
* Pain Numeric Scale
* Quebec questionnaire
* HAD questionnaire
* Blood samples for laboratory tests
* Randomization
* Proposal of the trial of virtual reality and collection of the informed consent, signed

Intervention protocol for patients randomized to Arm "virtual reality":

* Duration: 4 weeks
* 3 sessions per week of virtual reality (17 minutes of immersion and 15 minutes of rest)
* At each session: monitoring of heart rate during periods of rest and immersion) and control of blood pressure at the beginning and end of session.

M1 - 1 Month Visit

* Physical examination
* Pain Numeric Scale
* Quebec questionnaire
* HAD questionnaire
* Blood samples for laboratory tests M2 - 2 Month Visit
* Pain Numeric Scale
* Quebec questionnaire M3 - 3 Month Visit
* Pain Numeric Scale
* Quebec questionnaire M4 - 4 Month Visit
* Pain Numeric Scale
* Quebec questionnaire
* HAD questionnaire

ELIGIBILITY:
Inclusion Criteria:

* More than 18 and less than 60 years (inclusive)
* Chronic low back pain or chronic sciatica (between 3 months and 1 year of the current episode), without neurological deficit (low back pain more important than sciatica), common spinal origin, resistant to medical therapy, and the numerical pain scale > 30/100
* Written informed consent
* Membership or beneficiary of an insurance

Exclusion Criteria:

* Low back pain related to a spinal infectious disease, inflammatory, neoplasia, osteodystrophic, malformative and traumatic.
* Deficit sciatica (motor weakness and / or sensory)
* Low back pain secondary to failure of spinal intervention.
* Co-existence of pain of another etiology.
* Seizures.
* Psychiatric disorder, uncontrolled.
* Visual disturbances (significant decrease in visual acuity without correction possibility, problems with re-cognition of color, visual field loss).
* Inclusion in another trial to evaluate new ways of treating pain
* Sick leave over 1 year
* Pregnant women
* Inability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Low back pain in the last 48 hours | 4 months
  Low back pain in the last 48 hours assessed on a numerical pain scale (0 - 100) at 4 months

SECONDARY OUTCOMES:
Disability (Quebec questionnaire) | 1 month and 4 months
  Evaluation by quality of life questionnaries
Anxiety and depression (HAD) | 1 month and 4 months
  Evaluation by specific anxiety and depression questionnaries
Quality of life (SF-12) | at 1 and 4 months
  Evaluation by quality of life questionnaries
Overall serum antioxidant defenses | at inclusion (baseline) and 1 month after inclusion
  Determination of AOPP and carbonyl compounds, markers of oxidative stress and the TAS (total antioxidant status) that assesses the overall serum antioxidant defenses

CONTACTS AND LOCATIONS:
Overall Officials: Serge POIRAUDEAU, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France